CLINICAL TRIAL: NCT03563534
Title: Post-operative Pain After Silver Diamine Fluoride Application in Primary Molars With Deep Caries Versus Interim Restorative Therapy
Brief Title: Treatment of Primary Molars With Deep Caries Using Silver Diamine Fluoride
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manar Motawie Abdulfattah, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-06-44
Record Dates: First submitted 2018-06-10; First posted 2018-06-20 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Deep Caries
Keywords: Silver diamine fluoride, dental caries children
MeSH Terms: interventions — silver diamine fluoride; glass ionomer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- silver diamine fluoride (Active Comparator): 38% silver diamine fluoride applied to cavitated primary molars twice per week to arrest caries
  Interventions: Drug: Silver Diamine Fluoride
- interim restorative therapy (Active Comparator): Resin modified glass ionomer applied to cavitated primary molars
  Interventions: Drug: Glass Ionomer

INTERVENTIONS:
Drug: Silver Diamine Fluoride — Margins of cavitated lesion(s) will be excavated.The carious teeth will be isolated, kept dry, and apply 38% silver diamine fluoride.
  Arms: silver diamine fluoride
Drug: Glass Ionomer — Margins of cavitated lesion(s) will be excavated.The carious teeth will be isolated, kept dry, apply resin modified glass ionomer.
  Arms: interim restorative therapy

SUMMARY:
Untreated dental caries is a worldwide pandemic (Edelstein, 2006). Due to limited financial resources, poor access to basic oral care, and the high cost of restorative treatment, children of low-income nations have their general health, social well-being, and education opportunities affected by untreated dental caries (Baelum et al., 2007).

Traditional treatment of cavitated dentin lesions advocates complete removal of the decayed structure, i.e. the infected and affected dentin layers. During this procedure, however, a significant quantity of the dental structure is removed, and the pulp tissue may be exposed. In light of this, the complete removal of all decayed structures from a tooth with cavitated lesions is no longer seen as mandatory, as this increases the chance of pulp exposure, post-operative pain and weakens the tooth structure, and there is growing evidence to support incomplete removal of decayed tissue prior to the restoration of the cavity. It is argued, however, that carious lesions remaining in the cavity must be completely sealed in order to prevent their progression (Yee et al., 2009).

Arresting Caries Treatment (ACT) has been proposed to oversee untreated dental caries in children of disadvantaged communities. Treatment of carious lesions based on minimally invasive technique methods aim to prevent their progression and preserve pulp vitality by means of standards of anticipation, remineralization and minimal intervention in the dental tissue (Bedi and Sardo-Infirri, 1999).

DETAILED DESCRIPTION:
A treatment option has been proposed in the last decade, based on the change in understanding of carious biofilm development and caries progression. Sealing carious dentine beneath a restoration deprives the caries biofilm of nutrients and alters the environment sufficiently to slow or arrest lesion progression. This has the added benefit of avoiding pulp exposure and subsequent treatment (Santamaria, Innes, Machiulskiene, Evans, & Splieth, 2014).

There is no clear evidence that leaving soft infected dentine, before sealing the cavity, is deleterious. Instead, this may prevent pulp exposure, preserve the pulp vitality, reduce the permeability of the remaining dentine by stimulating tertiary dentine formation, and so change the environment for the remaining microorganisms and thus arresting caries process. Silver diamine fluoride (SDF), Ag(NH3)2F, has been used to arrest caries since 1969.Silver Diamine Fluoride is a topical drug that is applied clinically to control active dental caries and prevent further progression of disease. Although, the ideal way to treat teeth with decay is removal of the decay and placing a restoration, this alternative treatment allows us to stop decay with non-invasive methods, especially with young children that have primary teeth. Treatment with Silver Diamine Fluoride does not eliminate the need for restorative dentistry to repair function or aesthetics, but has been effective at prevention of further decay.

ELIGIBILITY:
Inclusion Criteria:

* CHILDREN

  * Aged 4 to 6 years.
  * in good general health.
* TEETH

  o Have at least one active dentin carious lesion on the occlusal surface of primary molars corresponding to ICDAS* codes 5 or 6*.
* PREOPERATIVE RADIOGRAPH

  * Absence of periapical infection.
  * No root resorption.
  * Normal periodontal ligament space.

Exclusion Criteria:

* CHILDREN

  * With systemic or neurological diseases.
  * With a history of allergy to silver or any substance present in the different materials to be used for treatment.
  * Unable to attend follow-up visits. TEETH
* With spontaneous pain, mobility or radiographic signs of pulpal or periapical infection.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Absence of spontaneous pain (questionnaire) | 6 months
  Direct questioning (yes/no)

SECONDARY OUTCOMES:
Absence of pain on percussion (clinical examination) | 6 months
  Applying pressure by finger (yes/no)
Absence of swelling (clinical examination) | 6 months
  Visual examination (yes/no)
periapical radiograph | 6 months
  absence of periapical radiolucency

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Al Manyal, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided